CLINICAL TRIAL: NCT05228431
Title: Single Arm and Phase II Clinical Trial of a Sandwich Regimen as XELOX Regimen and Capecitabine Alternate Administration Combined With Preoperative Intensity Modulated Radiation Therapy for pMMR Locally Advanced Rectal Cancer
Brief Title: Modified Sandwich Therapeutic Regimen for Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhen-Hai Lu (Other)
Responsible Party: Sponsor-Investigator, Zhen-Hai Lu, Pofessor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-494-Department of CRC
Record Dates: First submitted 2022-01-22; First posted 2022-02-08 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Advanced Rectal Cancer
Keywords: Rectal cancer; neoadjuvant chemoradiotherapy; optimization
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sandwich Regimen (Experimental): All rectal patients in this group will receive standard surgical resection.
  Interventions: Drug: XELOX; Drug: Capecitabine monotherapy; Radiation: Radiation

INTERVENTIONS:
Drug: XELOX — Starting from the first day of radiotherapy (set as day 0), the patient received a total of 4 courses of XELOX chemotherapy on days -42, -21, 42, and 63, including oxaliplatin 130 mg/m2, intravenous administration, d1, repeat every 3 weeks; and capecitabine 1000mg/m2, twice daily, d1-d14, repeat every 3 weeks.
Drug: Capecitabine monotherapy — During radiotherapy (Monday to Friday), capecitabine was administered at 1650 mg/m2/d, twice a day.
Radiation: Radiation — The TV is expanded by 6-7mm to form PTV1, and the CTV is expanded by 6-7mm to form PTV2. The dose of PTV1 was 50Gy/25 times/35 days, and the dose of PTV2 was 45Gy/25 times/35 days, 5 times/week for a total of 5 weeks.

SUMMARY:
In the treatment of locally advanced rectal cancer, the short-term and long-term efficacy of the traditional sandwich regimen has not reached satisfactory efficacy. For this reason, the concept of reducing the dose of postoperative chemotherapy or directly moving forward the full amount of postoperative chemotherapy was proposed, which is called total neoadjuvant therapy (TNT). However, TNT also includes the high toxicity of oxaliplatin in the whole process and the long time interval between the end of radiotherapy and the operation, which leads to fibrosis of the surrounding tissue, which increases the difficulty of surgical resection and makes it difficult to ensure good surgical specimen quality. In addition to this, there are issues that may increase the risk of potential disease progression in patients with poor treatment withdrawal. Therefore, appropriately reducing the intensity of chemotherapy and controlling the total duration of preoperative neoadjuvant therapy during radiotherapy is expected to alleviate the side effects of neoadjuvant therapy. Here, the investigators synthesized the characteristics of TNT and sandwich regimens and proposed a XELOX regimen and capecitabine alternate administration combined with preoperative intensity modulated radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

Pathological confirmed rectal adenocarcinoma.

Clinical stage T3-4 or T any N1.With or without MRF positivity, with or without EMVI positivity, R0 resection is estimated.

No metastasis

No signs of intestinal obstruction; or intestinal obstruction has been relieved after proximal colostomy surgery.

Age ranged from 18 to 75

No previous radiotherapy，surgery and chemotherapy.

Exclusion Criteria:

Multiple primary tumor

Cachexy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of pCR | One week after surgery
  rate of pathological complete remission

SECONDARY OUTCOMES:
DFS | 3 years
  Disease free survival
OS | 5 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Zhenhai Lu, Guangzhou, Guangdong, China